CLINICAL TRIAL: NCT06530186
Title: Evaluation of a Postcoital Sponge on Self-Reported Vaginal Health Parameters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Michael Ingber, Attending Physician, Atlantic Health System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AC-005
Record Dates: First submitted 2024-07-27; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Vaginal Infection; Vaginal Discharge; Vaginosis; Sexual Dysfunction
Keywords: vaginal odor; vaginal discharge; postcoital dripping; vaginal microbiome
MeSH Terms: conditions — Vaginitis; Vaginal Discharge; Vaginal Diseases; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- pH subset (Experimental): This subset of patients (n=100) will be checking their vaginal pH at various time intervals (before, 2-6 hours after, and 10-14 hours after sex).
  Interventions: Device: LiviWell Postcoital Vaginal Insert
- Main Cohort (Experimental): This subset of patients (n=900) will be providing user feedback on the study device, and will not be checking their vaginal pH
  Interventions: Device: LiviWell Postcoital Vaginal Insert

INTERVENTIONS:
Device: LiviWell Postcoital Vaginal Insert — subjects will use Livi within minutes of completion of sex, and will remove study device in under an hour.
  Other Names: Livi

SUMMARY:
LiviWell has developed a product designed for postcoital semen absorption. Previous studies have demonstrated the product rapidly absorbs semen, and leads to less symptoms of postcoital vaginal microbiome disruption such as vaginal odor and discharge. This study will investigate the study device, Livi, in a broader clinical setting.

DETAILED DESCRIPTION:
LiviWell's consumer hygiene device is a post-coital vaginal insert called "Livi". Livi is comprised of an applicator, with a medical-grade polyurethane foam and retrieval string. It is designed to be inserted into the vagina after intercourse to absorb semen deposited into the vaginal canal. The result is a decrease in discharge/dripping and vaginal odor. The investigators also believe the device will lower vaginal pH, as the typical premenopausal vaginal pH is acidic (pH ~4), and semen has an alkaline pH (~8). The resulting pH imbalance in sexually-active women not using male condoms had been shown to lead to vaginal odor, dripping, discomfort. Furthermore, the risk of bacterial vaginosis (BV) is higher in women who are sexually active and not using male condoms. The investigators have additional studies planned to evaluate if the product lowers the risk of BV.

The current study will be used to validate user needs requirements for the study device, understand pH changes after insertion, and evaluate change in symptoms of vaginal odor, discharge/dripping, and discomfort, common symptoms of vaginal microbiome disruption and bacterial vaginosis.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 (for pH subset, 18-45)
* Sexually-active with biological men
* Willing and able to use product
* Resides in continental USA
* Understands, reads, writes, and speaks English

Exclusion Criteria:

* Currently Pregnant or are trying to conceive
* Unable to use device due to poor motor function
* Unable to sign informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — No. Subjects must be biological females at birth in order to participate
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
User Experience Questionnaire | 24 hours
  Validation of User Needs Requirements as well as patient experience

SECONDARY OUTCOMES:
change in vaginal pH | 2-6 hours, and 10-14 hours after use
  change in vaginal pH before and after using Livi, and before and after NOT using Livi

CONTACTS AND LOCATIONS:
Locations (1):
- Garden State Urology, Mountain Lakes, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No